CLINICAL TRIAL: NCT00659516
Title: Smart Capnography Respiratory Index: Clinical Evaluation
Brief Title: Smart Capnography Respiratory Index in Post Anesthesia Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Rachel Weissbrod, Oridion Medical 1987 Ltd
Other Study IDs: 123
Record Dates: First submitted 2008-04-14; First posted 2008-04-16 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2008-04

CONDITIONS: Patients After Surgery and Anesthesia Monitored in the PACU

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: intubated patients
- 2: non intubated patients

SUMMARY:
The smart capnography respiratory index is a software tool that constitutes a representation of 4 parameters: End Tidal CO2, respiratory rate, O2 saturation and heart rate already displayed on a monitor in the form of a single respiratory index integer value ranging from 1 to 10 with trend information. The index is to be used to identify and display status and changes in patient respiratory status in a simple manner based on the summary of changes in the 4-above mentioned parameters. the respiratory index is to be used in varied clinical environments and is intended for use in adult and pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult or pediatric patients after surgery and anesthesia, monitored in the PACU

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the respiratory index evaluation will be performed on 40 patients (adult and pediatric) of which 30 will be non intubated
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-08 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
To demonstrate that the displayed respiratory index values and their associated description match the clinical status of the patients | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yaacov Gozal, MD, Principal Investigator — Shaare Zedek Medical center Jerusalem, Israel
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel